CLINICAL TRIAL: NCT04887480
Title: Direct Resuscitation of the Open Peritoneum: A Randomized Controlled Trial in Non-Traumatic Patients
Brief Title: Direct Resuscitation of the Open Peritoneum
Acronym: SH DROP
Status: Suspended | Phase: Not Applicable | Type: Interventional
Why Stopped: Funding paused
Sponsor: Sanford Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SH Ahmeti DROP Study
Record Dates: First submitted 2021-05-05; First posted 2021-05-14 (Actual); Last update posted 2024-01-19 (Actual); Status verified 2024-01

CONDITIONS: Wound; Abdomen; Abdomen, Acute; Wound Surgical
MeSH Terms: conditions — Abdominal Injuries; Abdomen, Acute; Surgical Wound | interventions — Glucose

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Negative Wound Pressure Therapy (Active Comparator): Negative Pressure Would Therapy
  Interventions: Device: Abthera™ Open Abdomen Negative Pressure Therapy Device System
- Negative Wound Pressure Therapy with Direct Peritoneal Resuscitation (Active Comparator): Negative Wound Pressure Therapy with Direct Peritoneal Resuscitation
  Interventions: Device: Abthera™ Open Abdomen Negative Pressure Therapy Device System; Drug: Dianeal PD-2 with 2.5% Dextrose

INTERVENTIONS:
Device: Abthera™ Open Abdomen Negative Pressure Therapy Device System — Suction set at -125mmHg
Drug: Dianeal PD-2 with 2.5% Dextrose — 800mL to 1000mL of Dianeal PD-2 into Abthera™ and dwell for 1 hour.
  Arms: Negative Wound Pressure Therapy with Direct Peritoneal Resuscitation

SUMMARY:
The DROP trial evaluates two ways of treating patients whose abdomens are left open after their abdominal surgery. The current standard of care at Sanford is for patients to have their wound covered with a sterile dressing connected to a vacuum with suction, which removes fluid from the abdomen. In this trial, we are evaluating the benefits of adding dialysis fluid to the abdomen periodically, prior to suctioning it out with the vacuum system. This trial will show if the addition of this fluid lowers the risk of complications and death, and allows the surgeon to close the abdomen sooner

ELIGIBILITY:
Inclusion Criteria:

* ≥18 years of age
* Have index operation performed by one of the Trauma and Acute Care surgeons at Sanford Medical Center Fargo
* Require an open abdomen due to a non-traumatic cause and placement of an Abthera™ wound vacuum
* Cognitively impaired adults will be included if a Legally Authorized Representative is available to provide informed consent.

Exclusion Criteria:

* Patients under the age of 18
* Vulnerable populations such as pregnant women and prisoners
* Patients with open abdomens as the result of trauma
* Non-English speaking (Due to time constraints pre-operatively and the length of time necessary to secure translation services, non-English speaking patients will not be enrolled).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2021-05-14 (Actual); Primary Completion 2025-05-30 (Estimated); Study Completion 2026-05-30 (Estimated)

PRIMARY OUTCOMES:
Major Complications | Through study completion, an average of 6 months
  Major complications (yes/no). Major complications include intra-abdominal abscess, wound dehiscence, anastomotic leak, intra-abdominal bleed, biloma, enterocutaneous fistula, evisceration, acute respiratory distress syndrome (ARDS)
Number of operations and time to closure | up to 4 weeks
  how many procedures/how long did it take to close the abdomen

SECONDARY OUTCOMES:
Length of ICU Stay | up to 4 weeks
  How many days was patient in ICU
Time on Vasopressors | up to 4 weeks
  How many days was patient on vasopressors

CONTACTS AND LOCATIONS:
Overall Officials: Mentor Ahmeti, MD, Principal Investigator — Sanford Health
Locations (1):
- Sanford Medical Center Fargo, Fargo, North Dakota, United States

IPD SHARING:
Plan to Share IPD: No